CLINICAL TRIAL: NCT01492283
Title: Pathophysiological Implications of the Incretin Hormones in Patients With Liver Disease With and Without Diabetes
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Jonatan I Bagger, MD PhD-student, University Hospital, Gentofte, Copenhagen
Other Study IDs: LINK-1-2011; H-1-2011-082 (Other: The Danish National Committee on Biomedical Research Ethics)
Record Dates: First submitted 2011-12-05; First posted 2011-12-14 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Non Alcoholic Fatty Liver Disease; Type 2 Diabetes; Liver Cirrhosis
Keywords: NAFLD; Incretin hormones
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Liver Cirrhosis | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA (whole blood) will be kept for 15 years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- NAFLD: Non alcoholic fatty liver disease without type 2 diabetes
  Interventions: Other: OGTT; Other: IIGI
- NAFLD+T2D: Non alcoholic fatty liver disease with type 2 diabetes
  Interventions: Other: OGTT; Other: IIGI
- T2D: Type 2 diabetics without non alcoholic fatty liver disease
  Interventions: Other: OGTT; Other: IIGI
- cirrhosis: Patients with liver cirrhosis
  Interventions: Other: OGTT; Other: IIGI
- Kontrol groups: Healthy control subjects
  Interventions: Other: OGTT; Other: IIGI

INTERVENTIONS:
Other: OGTT — 50g waterfree glucose dissolved in 300 ml water consumed over 5 min.
  Other Names: Waterfree glucose, The Pharmacy of the capital region
Other: IIGI — iso glycemic intravenous (iv) glucose infusion (IIGI) with 20% glucose
  Other Names: Glucose infusion, 20%

SUMMARY:
The main objective of this study is to analyze the pathophysiological implications of glucagon and the incretin hormones in patients with liver disease (Non alcoholic fatty liver disease (NAFLD) or cirrhosis) with and without diabetes compared with healthy controls. The present study will contribute significantly to the understanding of the pathophysiology of liver disease and glucose metabolism. The final goal is that the results could pave the way for new treatment modalities for patients with liver disease.

DETAILED DESCRIPTION:
Comparison of of insulin secretion (Area Under the Curve (AUC)) during the experimental days. Furthermore a comparison of GIP, GLP1 and glucagon responses as well as plasma glucose levels.

ELIGIBILITY:
I) Group 1: NAFLD patients with normal glucose tolerance Inclusion criteria

* NAFLD verified by a liver biopsy
* Caucasian >18 years of age
* Negative islet cell (ICA) and glutamic acid decarboxylase 65 (GAD65) autoantibodies
* Normal 75-g OGTT as specified in the WHO Criteria
* Normal haemoglobin and blood pressure (BP)
* Written informed consent

II) Group 2: NAFLD patients with type 2 diabetes Inclusion criteria

* NAFLD verified by liver biopsy
* T2DM according to the WHO Criteria
* Caucasian >18 years of age
* Negative ICA and GAD65, normal haemoglobin, normal BP
* Written informed consent

III) Group 3: NAFLD patients without type 2 diabetes Inclusion criteria

* NAFLD verified by liver biopsy
* Caucasian >18 years of age
* Normal 75-g OGTT
* Negative ICA and GAD65-autoantibodies
* Normal haemoglobin and BP
* Written informed consent

IV) Group 4: Cirrhosis with or without type 2 diabetes Inclusion criteria

* Liver cirrhosis verified by liver biopsy
* Caucasian > 18 years of age
* Negative ICA and GAD65-autoantibodies
* Normal haemoglobin and BP
* Written informed consent

V) Group 5: Healthy controls Inclusion criteria

* Caucasian >18 years of age
* Normal 75-g OGTT according to the WHO Criteria
* Negative ICA and GAD65-autoantibodies
* Normal haemoglobin and BP
* Written informed consent

Exclusion criteria (all groups)

* Other known liver disease - viral hepatitis, hereditary haemochromatosis, autoimmune liver disease, alpha-1 trypsin deficiency, Wilson disease, drug induced liver Injury (DILI)
* Treatment with medications that cannot be discontinued for 12 hours
* Unwillingness to participate in protocols
* Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with NAFLD and liver cirrhosis confirmed by liver biopsy, and patients with or without well characterized type 2 diabetes recruited in the the hospitals out patients clinic
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The Incretin effect | pre dose 0,10, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 240 min post dose
  The difference in insulin responses, as assessed by the area under curve (AUC) for plasma insulin and C-peptide concentrations, during the two different glucose stimuli: Oral glucose tolerance test (OGTT) and isoglycemic iv glucose infusion in NAFLD patients with and without diabetes, and cirrhotic patients compared to healthy control subjects

SECONDARY OUTCOMES:
Plasma Glucagon like peptide 1 (GLP-1) response | pre dose 0,10, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 240 min post dose
  Comparing GLP-1 responses of the different experimental days, compared to healthy control subjects.
Plasma Glucose-dependent insulinotropic peptide (GIP) response | pre dose 0,10, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 240 min post dose
  Comparing GIP responses of the different experimental days, compared to healthy control subjects.
Plasma glucagon response | pre dose 0,10, 20, 30, 40, 50, 60, 75, 90, 120, 150, 180, 240 min post dose
  Comparing glucagon responses of the different experimental days, compared to healthy control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Anders E Junker, MD, phd-student, Principal Investigator — Diabetes Research Division, Gentofte Hospital, University of Copenhagen
Locations (1):
- Diabetes Research Division, Gentofte University Hospital, Niels Andersens Vej 65, opgang 4b, 1. sal, Hellerup, Denmark

REFERENCES:
- [Derived] Lauritsen JV, Bergmann N, Junker AE, Gyldenlove M, Skov L, Gluud LL, Hartmann B, Holst JJ, Vilsboll T, Knop FK. Oral glucose has little or no effect on appetite and satiety sensations despite a significant gastrointestinal response. Eur J Endocrinol. 2023 Dec 6;189(6):619-626. doi: 10.1093/ejendo/lvad161. PMID 38035766
- [Derived] Maagensen H, Junker AE, Jorgensen NR, Gluud LL, Knop FK, Vilsboll T. Bone Turnover Markers in Patients With Nonalcoholic Fatty Liver Disease and/or Type 2 Diabetes During Oral Glucose and Isoglycemic Intravenous Glucose. J Clin Endocrinol Metab. 2018 May 1;103(5):2042-2049. doi: 10.1210/jc.2018-00176. PMID 29506157